CLINICAL TRIAL: NCT06748989
Title: Effect of a Specially Formulated Dietary Supplement With Pyrroloquinoline Quinone, γ-aminobutyric Acid, Caffeine and B-vitamins on Cognitive Function in Healthy Postmenopausal Women: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Cognitive Effects of a Dietary Supplement With PQQ, GABA, Caffeine, and B-Vitamins in Healthy Postmenopausal Women: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: FEMPHARMA Kft. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025CORTEXIUM
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Function and Memory

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participant will receive matching placebo supplement daily over a period of 6 weeks.
  Interventions: Dietary Supplement: Placebo food supplement
- Treatment (Experimental): Participants will receive Cortexium (a specially formulated dietary supplement with pyrroloquinoline quinone, γ-aminobutyric acid and B vitamins).
  Interventions: Dietary Supplement: Cortexium food supplement

INTERVENTIONS:
Dietary Supplement: Cortexium food supplement — Cortexium (a specially formulated dietary supplement with pyrroloquinoline quinone, γ-aminobutyric acid and B vitamins).
  Arms: Treatment
Dietary Supplement: Placebo food supplement — Placebo food supplement is completely identical weight and outlook capsule to Cortexium, with 50% microcrystalline cellulose and 50% starch.
  Arms: Placebo

SUMMARY:
Various food supplements have been shown to improve cognitive function. However, there is limited data on the impact of these supplements on postmenopausal women. Millions of women experience difficulty with concentration, and memory lapses during menopause. Research shows that up to 60% of women report cognitive changes related to menopause, severely impacting their quality of life and professional performance. Women are significantly more likely to develop dementia and other cognitive dysfunction. The specially formulated Cortexium with four key ingredients aims to support cognitive function in women:

* PQQ (Pyrroloquinoline Quinone) is a redox coenzyme with high antioxidant potential and is considered to affect the brain function by increasing mitochondrial production and activation, nerve cell protection, and enhanced production of nerve growth factor.
* GABA (gamma-aminobutyric acid) is an important neurotransmitter that helps induce calm and relaxation in the brain. Its positive effects include reducing stress and anxiety, which promotes mental clarity and concentration, thus enhancing mental performance. Additionally, it can help combat fatigue by supporting restful sleep, which, in the long term, boosts brain function efficiency.
* B-VITAMINS (B1, B2, B3, B5, B6, B7, B9, B12) are essential for brain function and energy production. They support the synthesis of neurotransmitters that improve mood, memory, and concentration, and help combat stress and mental fatigue. Together, they contribute to protecting brain cells and maintaining cognitive performance.
* CAFFEINE: The stimulating and invigorating effects of caffeine on the brain and nervous system have been known for centuries. Caffeine is a mild psychostimulant with invigorating effects. It also alleviates symptoms of fatigue and enhances work capacity. Moreover, moderate amounts of caffeine are known to have a stimulating effect on the cerebrocortical fields responsible for thinking: it enhances mental activity, improves cognitive functions, and accelerates mental associations. In this way, caffeine's stimulating effect can also lead to an improved sense of well-being Our aim is test the hypothesis that Cortexium dietary supplement improves cognitive function in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Good general health.
* Education level at least completed elementary.
* Menopausal status with minimum 1 year from the last menstrual period and based on the criterion of follicle-stimulating hormone (FSH) level (FSH > 30 mlU/ml) or a history of bilateral oophorectomy.

Exclusion Criteria:

* Active cancerous disease within the period of 5 years before recruitment.
* Mental diseases in medical history, including depression.
* Addiction to drugs and alcohol.
* Symptoms of dementia or history of neurological treatment or neurocognitive disorder.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Neurocognition Index (NCI) | From enrollment to the end of treatment at 6 weeks.
  Neurocognition Index (NCI) as calculated by Cognitive functions using the diagnostic instrument Central Nervous System-Vital Signs (CNS-VS) computerized neuropsychological / neurocognitive test.

SECONDARY OUTCOMES:
Central Nervous System-Vital Signs (CNS-VS) | From enrollment to the end of treatment at 6 weeks.
  Central Nervous System-Vital Signs (CNS-VS) 11 items of the cognitive function domain score (composite memory, verbal memory, visual memory, psychomotor speed, reaction time, complex attention, cognitive flexibility, processing speed, executive function, simple attention, and motor speed).

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Secret Private Clinic, Debrecen, HB, Hungary